CLINICAL TRIAL: NCT02700009
Title: Dissemination of Computer-assisted Cognitive-behavior Therapy for Depression in Primary Care
Brief Title: Computer-assisted Cognitive-Behavior Therapy for Depression in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: University of Denver (Other); University of York (Other)
Responsible Party: Principal Investigator, Jesse H Wright, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.0640; R18HS024047 (AHRQ)
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-assisted CBT (CCBT) (Experimental): 12 weeks of CCBT for depression
  Interventions: Behavioral: Computer-assisted CBT (CCBT)
- Treatment as Usual (TAU) (Active Comparator): Treatment as usual by primary care physicians
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Computer-assisted CBT (CCBT) — Computer-assisted psychotherapy for depression using a computer program plus clinician support
  Arms: Computer-assisted CBT (CCBT)
Other: Treatment as Usual (TAU) — Ordinary treatment for depression in primary care setting
  Arms: Treatment as Usual (TAU)

SUMMARY:
Computer-assisted cognitive-behavior therapy, a treatment that has been shown to be effective in previous studies in psychiatric settings, will be disseminated into primary care - a health care setting where there are significant problems in receiving adequate treatment for depression. Computer-assisted cognitive-behavior therapy will feature a low-cost method of delivering therapy designed to be replicated and sustained in other primary care settings. Feasibility and effectiveness will be tested by randomly assigning 320 primary care patients with depression to receive either computer-assisted cognitive-behavior therapy or treatment as usual.

DETAILED DESCRIPTION:
Computer-assisted cognitive-behavior therapy (CCBT) for depression in primary care will be evaluated in a trial with 320 patients randomly assigned to CCBT or treatment as usual (TAU). The study will disseminate a therapy method found to be effective in psychiatric settings into primary care - a setting where there have been significant problems in delivery of adequate, evidence-based treatment for depression. The study will include a high percentage of disadvantaged patients - a population that has been largely ignored in previous research in CCBT. There have been no previous studies of CCBT for depression in primary care that have enrolled large numbers of disadvantaged patients. The form of CCBT used in this study is designed to increase access to effective therapy, provide a cost-effective method, and be a sustainable model for wide-spread use in primary care.

In order to deliver therapy in a practical manner that can be replicated in other primary care practices, patients with significant symptoms of depression will receive treatment with an empirically supported computer program that builds cognitive-behavior therapy skills. Support for CCBT will be provided by telephone and/or e-mail contact with a care coordinator instead of the face-to-face treatment with a cognitive-behavior therapist that has been a part of CCBT delivery in mental health settings. Novel features of this treatment program include: 1) fully detailed and replicable method for integrating clinician support with CCBT in primary care; 2) delivery of CCBT to a population with high percentage of disadvantaged patients; 3) integration of CCBT into the primary care delivery model; 4) highly interactive, multimedia computer program with adaptations for persons who may have lower levels of education or computer experience; 5) advanced cost-benefit analysis including data on actual health care utilization and costs; 6) exploration of moderators and predictors of treatment outcome.

Outcome will be assessed by measuring CCBT completion rate, comprehension of CBT concepts, and satisfaction with treatment; in addition to ratings of depressive symptoms, negative thoughts, and quality of life. The cost-effectiveness analysis and exploration of possible predictors of outcome should help clinicians, health care organizations, and others plan further dissemination of CCBT in primary care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Health Questionnaire score of 10 or above
2. Age 18 or above

Exclusion Criteria:

1. Refusal to provide informed consent
2. Inability to read English text on computer screen
3. Significant suicidal thoughts, intent, plan, or behavior reported on Columbia Suicide Severity Rating Scale
4. Severe or poorly controlled medical disorders that would interfere with participation in CCBT (e.g., liver failure, terminal cancer)
5. Dementia or other organic brain disorders that would prevent participation in CCBT
6. Diagnosis of any psychotic disorder or bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-05; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment period ends
  Self-report scale for depression

SECONDARY OUTCOMES:
Automatic Thoughts Questionnaire | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment period ends
  Self-report measure of negative cognitions
Quality of Life Enjoyment and Satisfaction Questionnaire | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment period ends
  Self-report measure of quality of life
Client Service Receipt Inventory | Change from baseline after 12 weeks of treatment and 3 and 6 months after 12-week treatment ends
  Record of medical and related services
Quality of Well Being Scale | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment periods ends
  Self-report measure of well-being
Patient Attitudes and Expectations Scale | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment periods ends
  Assessment of patient attitudes toward treatment
Generalized Anxiety Disorder - 7 | Change from baseline after 12 weeks of treatment and 3 and 6 months after the 12-week treatment period ends
  Self-report measure of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Wright, M.D., Ph.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, School of Medicine, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wright JH, Owen J, Eells TD, Antle B, Bishop LB, Girdler R, Harris LM, Wright RB, Wells MJ, Gopalraj R, Pendleton ME, Ali S. Effect of Computer-Assisted Cognitive Behavior Therapy vs Usual Care on Depression Among Adults in Primary Care: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2146716. doi: 10.1001/jamanetworkopen.2021.46716. PMID 35142833

DOCUMENTS (1):
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02700009/ICF_000.pdf